CLINICAL TRIAL: NCT06451393
Title: A Radio-Pathomic Multimodal Machine Learning Model for Predicting Pathological Complete Response to Neoadjuvant Chemotherapy in Advanced Gastric Cancer: A Retrospective Observational Study
Brief Title: Predicting Gastric Cancer Response to Chemo With Multimodal AI Model
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: E2021088
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Chemotherapy Effect
Keywords: Advanced gastric cancer; Neoadjuvant chemotherapy; Multimodal; Pathological complete response
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant chemotherapy with radical tumor resection surgery: (i) Patients with indistinguishable tumor lesions on the CT images due to insufficient filling of the stomach during the CT inspection; (ii) patients without indistinguishable tumor cell on the pathological slides due to inadequate sampling; (iii) patients with insufficient data.
  Interventions: Drug: Neoadjuvant chemotherapy with radical tumor resection surgery

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy with radical tumor resection surgery — All patients were pathologically diagnosed as advanced gastric cancer, all receive neoadjuvant chemotherapy, after the completion of neoadjuvant chemotherapy, all patients receive radical tumor resection surgery (partial gastrectomy or total gastrectomy, as proper).

SUMMARY:
This study aims to develop a multimodal model combining radiomic and pathomic features to predict pathological complete response (pCR) in advanced gastric cancer patients undergoing neoadjuvant chemotherapy (NAC). The researchers intended to collected pre-intervention CT images and pathological slides from patients, extract radiomic and pathomic features, and build a prediction model using machine learning algorithms. The model will be validated using a separate cohort of patients. This research intend to build a radiomic-pathomic model that can outperform models based on either radiomic or pathomic features alone, aiming to improve the prediction of pCR in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically confirmed adenocarcinoma of the stomach or esophagogastric junction who received NAC and radical gastrectomy;
* patients who underwent abdominal multidetector computed tomography (CT) inspection, gastroscope, and tumor tissue biopsy before any intervention started;
* Lesions that are assessable according to The Response Evaluation Criteria in Solid Tumors Version 1.1

Exclusion Criteria:

* Patients with indistinguishable tumor lesions on the CT images due to insufficient filling of the stomach during the CT inspection;
* patients without indistinguishable tumor cell on the pathological slides due to inadequate sampling;
* patients with insufficient data.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed adenocarcinoma of the stomach or esophagogastric junction who received neoadjuvant chemotherapy and radical gastrectomy;
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | Assessed within 30 days after radical resection surgery.
  Pathological complete response (pCR) was defined as no viable cells remained in the primary tumor lesions and the dissected lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Junsheng Peng, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from Dr. Junsheng Peng (E-mail: pengjsh@mail.sysu.edu.cn) upon reasonable request.